CLINICAL TRIAL: NCT06843434
Title: A Phase II Study of Neoadjuvant Botensilimab and Balstilimab Immunotherapy for Mismatch Repair Proficient Rectal Adenocarcinoma
Brief Title: A Study of Botensilimab and Balstilimab for Rectal Adenocarcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-389
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Microsatellite Stable Rectal Carcinoma; Locally Advanced Rectal Adenocarcinoma
Keywords: Microsatellite Stable Rectal Carcinoma; mismatch repair proficient locally advanced rectal adenocarcinoma; locally advanced rectal adenocarcinoma; microsatellite stable locally advanced rectal adenocarcinoma; Memorial Sloan Kettering Cancer Center; 24-389
MeSH Terms: interventions — balstilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Participants with locally advanced rectal cancer (Experimental): Up to 40 patients with mismatch repair proficient (MMRp)/microsatellite stable (MSS) locally advanced (stage II or III) rectal cancer
  Interventions: Drug: Balstilimab; Drug: Botensilimab

INTERVENTIONS:
Drug: Balstilimab — Balstilimab is a fully human monoclonal IgG4 antibody designed to block PD-1 binding to PD-L1 and PD-L2
Drug: Botensilimab — Botensilimab is a novel fully human fragment crystallizable (Fc)-engineered immunoglobulin 1 kappa (IgG1κ) anti-CTLA-4 immunoglobulin G1 (IgG1) antagonist antibody that is designed to optimally promote fragment-crystallizable gamma receptor (FcγR) effector functions that are important for enhancing T cell priming and regulatory T cell (Treg) depletion.

SUMMARY:
The purpose of this study is to find out whether the combination of botensilimab and balstilimab (BOT/BAL) is a safe and effective treatment that causes few or mild side effects for people with mismatch repair proficient (MMRp)/microsatellite stable (MSS) locally advanced rectal adenocarcinoma. The investigators will also find out whether BOT/BAL is an effective treatment when given in combination with standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for trial.

  a. If participant is unable to provide written informed consent, the legally authorized representative (LAR) of the person who is being asked to participate in this research study may give consent on the participant's behalf.
* Be ≥18 years of age on the date of signing informed consent.
* ECOG performance status of 0 or 1.
* Histologically confirmed rectal adenocarcinoma.
* Adenocarcinoma with distal margin of 15 cm or less from the anal verge on endoscopy, staged with endorectal ultrasound (ERUS) or magnetic resonance imaging (MRI) as cT3/cT4 N0 or cT(any) cN1/2.
* No evidence of distant metastases
* Radiologically measurable or clinically evaluable disease per Protocol Section 13.0.
* Tumor specimen that demonstrates intact mismatch repair enzymes by immunohistochemistry or microsatellite stability as demonstrated by NGS or PCR.
* Negative pregnancy test done within 14 days prior to beginning treatment, for women of childbearing potential only. Subjects of childbearing potential must be willing to use an adequate method of contraception. Appropriate methods of birth control include abstinence, oral contraceptives, implantable hormonal contraceptives, or double barrier method (diaphragm plus condom). Contraception is required for the course of the study starting with the first dose of study medication through 150 days after the last dose of study medication. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Nonchildbearing potential is defined as follows (by other than medical reasons):

  1. ≥45 years of age and has not had menses for >1 year
  2. Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  3. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study.
* Demonstrate adequate organ function as defined in the Table 6-1 below within 14 days of Cycle 1 Day 1, and all screening labs should be performed within 14 days of treatment initiation.

Hematological Absolute neutrophil count (ANC): ≥1,500 /mm^3 Platelets: ≥100,000 / mcL Hemoglobin: ≥8.0 g/dL

Renal Serum creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl): ≤1.5 × upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 × institutional ULN AST (SGOT) and ALT (SGPT): ≤ 2.5 × ULN

Coagulation International normalized ratio (INR) or Prothrombin time (PT) or activated partial thromboplastin time (aPTT): For patients not taking warfarin: INR ≤ 1.5 or PT ≤ 1.5 x ULN; and either PTT or aPTT ≤ 1.5 x ULN. Patients on warfarin may be included on a stable dose with a therapeutic INR <3.5

Exclusion Criteria:

* Recurrent rectal cancer.
* Prior pelvic radiation therapy, chemotherapy, or surgery for rectal cancer.
* Tumor is causing symptomatic bowel obstruction (patients who have a temporary diverting ostomy are eligible).
* Other invasive malignancy ≤ 2 years prior to registration. Exceptions are non-melanoma skin cancer that has undergone potentially curative therapy and in situ cervical carcinoma.
* Active infection requiring systemic therapy.
* Other anticancer or experimental therapy. No other experimental therapies (including chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, angiogenesis inhibitors, matrix metalloprotease inhibitors, thalidomide, anti-VEGF/Flk-1 monoclonal antibody or other experimental drugs) of any kind are permitted while the patient is receiving study treatment.
* Known history of interstitial lung diseases/pneumonitis
* Known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Known active hepatitis B (e.g., HbsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Live vaccination within 28 days prior to receiving the first dose of immunotherapy. The use of inactivated seasonal influenza vaccines (e.g., Fluzone®) will be permitted on study without restriction.
* Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine or booster < 7 days before C1D1. For vaccines requiring more than 1 dose, the full series should be completed prior to C1D1, when feasible. Booster shot not required but also must be administered > 7 days from C1D1 or > 7 days from future cycle on study
* Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke or myocardial infarction within 180 days of enrollment, unstable angina, congestive heart failure (New York Heart Association class ≥ III), or serious uncontrolled cardiac arrhythmia requiring medication.

  a. QTcF (QT interval corrected using Fridericia's formula) of ≥450 ms.
* Known active tuberculosis.
* Receiving systemic corticosteroid therapy 1 week prior to the first dose of study drug or receiving any other form of systemic immunosuppressive medication.

  a. Corticosteroid use as a premedication for IV contrast allergies/reactions is allowed. Subjects who are receiving daily corticosteroid replacement therapy are also an exception to this rule. Daily prednisone at doses of ≤ 7.5 mg or equivalent hydrocortisone dose are examples of permitted replacement therapy. Use of inhaled or topical corticosteroids is permitted.
* Has ongoing or recent (within 5 years) evidence of significant autoimmune disease or any other condition that required treatment with systemic immunosuppressive treatments. The following are not exclusionary: vitiligo, childhood asthma that has resolved, endocrinopathies (such as hypothyroidism or type 1 diabetes) that require only hormone replacement.
* Prior allogeneic tissue/solid organ transplant, except for corneal transplants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-20 (Actual); Primary Completion 2028-02-20 (Estimated); Study Completion 2028-02-20 (Estimated)

PRIMARY OUTCOMES:
Best Overall Response Rate | 1 year
  The primary objective of this study is to determine the best overall response rate (ORR) after initial neoadjuvant combination botensilimab and balstilimab in subjects with MMRp/MSS locally advanced (stage II or III) rectal adenocarcinoma. ORR is defined by rectal MRI and endoscopic exam and graded as progressive disease (PD), stable disease (SD) (sustained for 3 months), partial response (PR), near complete response (nCR) and clinical complete response (cCR). Patients with PR, nCR, or cCR will be considered responders, while the rest will be non-responders.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Cercek, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center at Suffolk - Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org